CLINICAL TRIAL: NCT05859724
Title: A Randomized, Double-blind, Placebo-controlled, Single- and Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, Pharmacodynamics and Exploratory Clinical Activity of NM26-2198 in Healthy Volunteers and in Adult Patients With Atopic Dermatitis
Brief Title: Evaluation of NM26-2198 in Healthy Subjects and in Patients With Moderate-to-severe Atopic Dermatitis (AD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Asset acquisition by Johnson & Johnson. Minimum study objectives necessary to inform safety, tolerability, and dose selection for Phase 2 dose-ranging evaluation of NM26-2198 were achieved, with full completion of all healthy volunteer cohorts.
Sponsor: Yellow Jersey Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB-NM026-2198-101; 2023-503577-38 (EudraCT Number)
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for NM26-2198) for subcutaneous (SC) injection in healthy volunteers (HVs) on Day 1 (SAD Cohorts) and on Days 1, 8, 15, and 22 (MAD Cohorts)
  Interventions: Other: Placebo
- NM26-2198 (Experimental): NM26-2198 10mg, 50mg, 150mg, 300mg, 400mg, 600mg, and 900mg for SC injection in HVs on Day 1 (SAD Part A); NM26-2198 150mg and 300mg for SC injection in patients with AD on Days 1, 8, 15, and 22 (MAD Part B); NM26-2198 150mg and 300mg for SC injection in HVs on Days 1, 8, 15, and 22 (MAD Part C)
  Interventions: Biological: NM26-2198

INTERVENTIONS:
Biological: NM26-2198 — IL-4R/IL-31 bispecific antibody for subcutaneous administration
  Arms: NM26-2198
Other: Placebo — Placebo for NM26-2198
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single- and multiple ascending dose study of subcutaneous (SC) administration of NM26-2198 in healthy volunteers and adult patients with moderate to-severe AD to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single (SAD) and multiple doses (MAD) of NM26-2198.

ELIGIBILITY:
Inclusion Criteria:

1. SAD: Non-Asian ethnicity with grandparents and parents of non-Asian descent or Japanese descent having all four Japanese grandparents born in Japan.
2. SAD and MAD in Healthy Volunteers: Male or female aged 18 to 55 years; MAD: Male or female ≥18 years of age.
3. ALL COHORTS: Weight of 45 kg to 100 kg and BMI of 18.0 to 30.0 kg/m2.
4. SAD and MAD in Healthy Volunteers: Non-childbearing, non-breastfeeding females or males willing to use double barrier contraception or abstention from sex and sperm donation during the study; MAD: Males willing to use double barrier contraception or abstention from sex and sperm donation during the study; non-childbearing females or females of childbearing potential using protocol-defined method contraception, and who is not pregnant, lactating, or breastfeeding.
5. MAD: Diagnosis of chronic AD.
6. MAD: EASI score ≥16.
7. MAD: vIGA-AD™ score of ≥3.
8. MAD: Atopic lesions cover ≥10% of body surface area (BSA).
9. MAD: PP-NRS score ≥4.
10. MAD: Daily use of non-prescription emollient.

Note: Other protocol-defined Inclusion criteria apply.

Exclusion Criteria:

1. SAD and MAD in Healthy Volunteers: Any clinically-relevant medical history or lab abnormality, including positive test for SARS-CoV-2, Hepatitis B or C, or HIV; MAD: Clinically-significant, abnormal laboratory findings, or positive test for SARS-CoV-2, Hepatitis B or C, or HIV.
2. ALL COHORTS: Clinically important ECG abnormalities or history/evidence thereof.
3. SAD and MAD in Healthy Volunteers: Use of prescription or non-prescription medications (except occasional use of paracetamol).
4. MAD: Diagnosis of protocol-specified skin diseases other than AD, or history of other significant skin condition that could interfere with study assessments.
5. MAD: History or ongoing allergy/hypersensitivity or history, or history of hypersensitivity to biological drugs.
6. MAD: Recent receipt of immunoglobulin or blood products.
7. MAD: Recent treatment with protocol-specified investigational treatments, or any prior treatment with dupilumab, tralokinumab, lebrikizumab, nemolizumab, or other protocol-specified drugs.
8. MAD: AD with recent ocular involvement requiring chronic ocular corticosteroid treatment.
9. MAD: Chronic pruritis due to conditions other than AD.
10. MAD: Acute AD superinfection, recent superficial skin infection, or other chronic/acute infection requiring protocol-defined treatments.
11. MAD: Recent use of sedating antihistimines, systemic corticosteroids, cytotoxic treatments, other immunosuppressive/immunomodulating agents, and other protocol-specified prohibited medications.
12. MAD: Recent topical corticosteroid or prescription moisturizer use.

Note: Other protocol-defined Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Treatment Emergent Adverse Events (TEAEs) [SAD] | First dose through end of study (Day 57)
  TEAEs defined as AEs and SAEs developing or worsening during treatment period (time from the first dose of study drug up to the end of study visit [Day 57 in SAD]), and includes findings from vital signs, electrocardiogram (ECG), clinical laboratory tests, physical examinations, and injection site evaluations.
Percentage of participants with Treatment Emergent Adverse Events (TEAEs) [MAD] | First dose through end of study (Day 85)
  TEAEs defined as AEs and SAEs developing or worsening during treatment period (time from the first dose of study drug up to the end of study visit [Day 85 in MAD]), and includes findings from vital signs, electrocardiogram (ECG), clinical laboratory tests, physical examinations, and injection site evaluations.

SECONDARY OUTCOMES:
Pharmacokinetics of NM26-2198: Peak Concentration (Cmax) [SAD] | Pre-dose on Day 1 through Day 57
  Mean maximum concentration of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Peak Concentration (Cmax) [MAD] | Pre-dose on Day 1 through Day 85
  Mean maximum concentration of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Trough Concentration (Ctrough) [MAD] | Pre-dose on Day 1 through Day 85
  Mean trough concentrations of NM26-2198 with multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Time of Peak Concentration (Tmax) [SAD] | Pre-dose on Day 1 through Day 57
  Mean time of maximum concentration of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Time of Peak Concentration (Tmax) [MAD] | Pre-dose on Day 1 through Day 85
  Mean time of maximum concentration of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Last Area Under the Curve (AUClast) [SAD] | Pre-dose on Day 1 through Day 57
  Mean area under the curve from the time of dosing to the last measurable concentration of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Last Area Under the Curve (AUClast) [MAD] | Pre-dose on Day 1 through Day 85
  Mean area under the curve from the time of dosing to the last measurable concentration of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Area Under the Curve During the Dosing Interval (AUCtau) [SAD] | Pre-dose on Day 1 through Day 7
  Mean area under concentration-time curve over dosing interval of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Area Under the Curve During the Dosing Interval (AUCtau) [MAD] | Pre-dose on Day 1 through Day 29
  Mean area under concentration-time curve over dosing interval of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Estimated Total Exposure (AUCinf) [SAD] | Pre-dose on Day 1 through Day 57
  Mean estimated total exposure to NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Estimated Total Exposure (AUCinf) [MAD] | Pre-dose on Day 1 through Day 85
  Mean estimated total exposure to NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Time-Averaged Concentration (AUC%extrap) [SAD] | Pre-dose on Day 1 through Day 57
  Mean time-averaged concentration of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Time-Averaged Concentration (AUC%extrap) [MAD] | Pre-dose on Day 1 through Day 85
  Mean time-averaged concentration of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Time of last quantifiable concentration (tlast) [SAD] | Pre-dose on Day 1 through Day 57
  Mean estimated time to last quantificable concentration of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Time of last quantifiable concentration (tlast) [MAD] | Pre-dose on Day 1 through Day 85
  Mean estimated time to last quantificable concentration of NM26-2198 after multiple dose administration in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Terminal Elimination Rate (λz) [SAD] | Pre-dose on Day 1 through Day 57
  Mean terminal elimination rate of NM26-2198 after single dose administrations in healthy subjects.
Pharmacokinetics of NM26-2198: Terminal Elimination Rate (λz) [MAD] | Pre-dose on Day 1 through Day 85
  Mean terminal elimination rate of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Terminal elimination half-life (t1/2) [SAD] | Pre-dose on Day 1 through Day 57
  Mean terminal elimination half-life of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Terminal elimination half-life (t1/2) [MAD] | Pre-dose on Day 1 through Day 85
  Mean terminal elimination half-life of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Total body clearance (CL/F) [SAD] | Day 1
  Mean total body clearance of NM26-2198 after single dose administration in healthy subjects.
Pharmacokinetics of NM26-2198: Total body clearance (CL/F) [MAD] | Day 1 and Day 22
  Mean total body clearance of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Apparent volume of distribution (Vz/F) [SAD] | Day 1
  Mean apparent volume of distribution of NM26-2198 after single dose administrations in healthy subjects.
Pharmacokinetics of NM26-2198: Apparent volume of distribution (Vz/F) [MAD] | Day 1 and Day 22
  Mean apparent volume of distribution of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Accumulation ratio of last dose Cmax (Racc,cmax) [MAD] | Day 1 through Day 22
  Mean accumulation ratio of last dose Cmax of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Pharmacokinetics of NM26-2198: Accumulation ratio of last dose AUCtau (Racc,AUCtau) [MAD] | Day 1 through Day 22
  Mean accumulation ratio of last dose AUCtau of NM26-2198 after multiple dose administrations in healthy volunteers and in patients with AD.
Percentage of subjects developing treatment-emergent anti-drug antibodies (ADAs) [SAD] | Pre-dose on Day 1 through Day 57
Percentage of subjects developing treatment-emergent anti-drug antibodies (ADAs) [MAD] | Pre-dose on Day 1 through Day 85
Percentage of subjects developing treatment-enhanced anti-drug antibodies (ADAs) [SAD] | Pre-dose on Day 1 through Day 57
Percentage of subjects developing treatment-enhanced anti-drug antibodies (ADAs) [MAD] | Pre-dose on Day 1 through Day 85
Mean ADA titers [SAD] | Pre-dose on Day 1 through Day 57
Mean ADA titers [MAD] | Pre-dose on Day 1 through Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Yellow Jersey Therapeutics AG Clinical trial, Study Director — Yellow Jersey Therapeutics AG
Locations (15):
- United States (6):
  - First OC Dermatology Research, Fountain Valley, California
  - California Clinical Trials Medical Group (CCTMG) managed by Parexel, Glendale, California
  - TCR Medical Corporation, San Diego, California
  - D&H Tamarac Research Center, Tamarac, Florida
  - Sadick Research Group, New York, New York
  - Paddington Testing Co., Philadelphia, Pennsylvania
- Canada (2):
  - DermEffects, London, Ontario
  - Centre de Recherche Saint-Louis, Québec
- Germany (3):
  - Universitätsmedizin Mainz, Mainz, Hesse
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - UK-SH - Lübeck, Lübeck, Schleswig-Holstein
- Poland (4):
  - COPERNICUS Podmiot Leczniczy Sp. z o.o., Szpital Sw. Wojciecha, Gdansk
  - Uniwersytecki Szpital Kliniczny im. F.Chopina w Rzeszowie, Rzeszów
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw

IPD SHARING:
Plan to Share IPD: No